CLINICAL TRIAL: NCT01300182
Title: The Effect of Early Whole-Body Vibration Therapy on Neuromuscular Control After Anterior Cruciate Ligament Reconstruction
Brief Title: The Effect of Early WBVT on Neuromuscular Control After ACLR
Acronym: WBVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fu Chak Lun Allan, Mr Fu Chak Lun Allan, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: wbvtrct
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: ACLR
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole body vibration therapy (Experimental): Whole body vibration therapy on top of conventional physiotherapy treatment.
  Interventions: Other: Whole body vibration therapy
- Control (Active Comparator): Conventional post-operative physical therapy rehabilitation exercises.
  Interventions: Other: Control

INTERVENTIONS:
Other: Whole body vibration therapy — The WBVT will be carried out in a vibration plates operated in vertical direction. The frequency of that vibration can be adjusted step of 5Hz with vibration frequency ranges from 20Hz to 60Hz. The amplitude can be set as 4mm.
  Other Names: Fitvibe Excel Pro - model number: 332015 (N.V. GymnaYniphy, Bilzen, Belgium)
  Arms: Whole body vibration therapy
Other: Control — Conventional post-operative physical therapy exercises and rehabilitation.
  Arms: Control

SUMMARY:
To investigate the effect of early WBVT on neuromuscular control after ACLR.

DETAILED DESCRIPTION:
The knee joint position sense, postural control, muscular strength and functional ability after anterior cruciate ligament construction (ACLR) are distorted, and even after a period of rehabilitation.

Previous studies had demonstrated that there was improvement in knee joint, postural balance, muscle strength and functional outcome in elderly, stroke and spastic patients already. It has also been concluded that the balance in elderly, postmenopausal women, Parkinson's disease, multiple sclerosis, stroke and spastic patients were all significantly improved. Some studies showed that the proprioception in osteoarthritis patients significantly improve. Knee strength is also one of the aspect being improved.

However, no studies focus on the early effect of WBVT on knee joint proprioception, postural control, muscle strength, knee joint stability and functional ability in ACLR cases. This study is to answer this research gap.

ELIGIBILITY:
Inclusion Criteria:

* ACLR with a single-bundle approach
* no complication such as wound infection after the ACLR
* able to walk with a pair of elbow crutches independently at one month post operation

Exclusion Criteria:

* concomitant posterior cruciate ligament, lateral collateral ligament, and medial collateral ligament injury in the same knee
* previous operation on either lower limbs
* medical problems such as pregnancy, acute thrombosis, serious cardiovascular disease, pacemaker, acute hernia, discopathy, spondylolysis, severe diabetes, epilepsy, recent infections, severe migraine, tumors or kidney stones etc
* neurological conditions such as Guillain-Barre ́ syndrome, myasthenia gravis, and postpolio syndrome
* prior experience of WBVT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Joint position sense | 1-month post-operation, 3-months post-operation, 6-months post-operation
  Using Biodex Dynamometer (Biodex Medical Systems, Shirley, NY, USA) for measurement.
Muscle isokinetic strength | Pre-operation, 3-months post-operation, 6-months post-operation
  Using Cybex NORM dynamometer for measurement.
Postural control | 1-month post-operation, 3-months post-operation, 6-months post-operation
  Using Biodex Stability System (BSS; Biodex Medical Systems, Shirley, NY, USA with software version 3.1) for measurement
Functional Outcome | Pre-operation and 6-months post-operation
  Functional Outcomes
  * single leg hop test
  * triple leg hop test
  * caricoca test
  * Shuttle run test
Knee joint stability | Pre-operation, 3-months post-operation, 6-months post-operation
Knee range of motion | 6-months post operation

CONTACTS AND LOCATIONS:
Overall Officials: Chak Lun Allan Fu, Principal Investigator — Physiotherapy Department, Prince of Wales Hospital
Locations (1):
- Physiotherapy Department, Prince of Wales Hospital, Shatin, Hong Kong, Hong Kong